CLINICAL TRIAL: NCT06793332
Title: Prospective, One-arm, Phase II Clinical Study of Ivoximab Combined with TROP2 ADC in the Treatment of Brain Metastases in Triple-negative Breast Cancer
Brief Title: BrAin Metastasis in TripLe Negateive Breast Cancer: IvoneScimab and Trop2 ADC
Acronym: BALISTA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Director of Phase I clinical Research ward, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BALISTA（YBCSG-24-01）
Record Dates: First submitted 2024-12-28; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Triple-Negative Breast Cancer (TNBC); Brain Metastases
Keywords: triple-negative breast cancer; brain metastases; Ivonescimab; TROP2 ADCs
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ivonescimab combined with TROP2 ADC (Experimental)
  Interventions: Drug: Ivonescimab Combined With TROP2 ADC

INTERVENTIONS:
Drug: Ivonescimab Combined With TROP2 ADC — Ivonescimab: 20 mg/kg, ivggt, day 1, every 3 weeks; Sacituzumab govitecan: 10 mg/kg, ivggt, day 1 and day 8, every 3 weeks;
  Other Names: AK112 Combined With TROP2 ADC

SUMMARY:
This study is a single-center, prospective, single-arm clinical trial, which intends to enroll patients with triple-negative breast cancer with brain metastases to receive ivonescimab combined with TROP2 ADC (such as sacituzumab govitecan) treatment until disease progression, intolerable toxicity, withdrawal of informed consent, or the investigator deems it necessary to discontinue the medication, and to collect data on the drug's efficacy and safety.

DETAILED DESCRIPTION:
Brain metastasis is a common site of metastasis in triple-negative breast cancer (TNBC), with an incidence rate of approximately 30-45%. Once breast cancer patients develop brain metastasis, their survival period is short and prognosis is poor. The median overall survival (mOS) of TNBC patients with brain metastasis is even less than 6 months. Therefore, it is necessary and urgent to explore effective treatment regimens to improve the survival of patients with breast cancer brain metastasis.

In recent years, several novel drugs, including immunotherapy, anti-angiogenic targeted therapy, and antibody-drug conjugates (ADCs), have achieved significant success in metastatic TNBC, significantly improving the prognosis and survival of advanced TNBC. The combination of immune checkpoint inhibitors and anti-angiogenic therapy has also become an important treatment strategy for TNBC. The results of a phase Ib/II study of PM8002 (a bispecific antibody targeting PD-L1 and VEGF-A, exerting both immune and anti-angiogenic effects) combined with albumin-bound paclitaxel in the treatment of advanced TNBC patients showed that the objective response rate (ORR) was 78.6%, and the median progression-free survival (mPFS) was 14 months. AK112, a bispecific antibody targeting PD-1 and VEGF-A, combined with chemotherapy, was approved by the National Medical Products Administration（NMPA） of Cnina on May 10, 2024, for the treatment of patients with advanced non-squamous NSCLC with EGFR mutations who have progressed after EGFR-TKI treatment. Notably, the efficacy analysis of NSCLC patients with baseline brain metastasis in the 201/202 studies of AK112 showed that the intracranial response rate of AK112 combined with platinum-based chemotherapy was 39% (including 25% complete response); the intracranial response rate of AK112 monotherapy also reached 14%. For untreated brain metastasis patients, the intracranial mPFS of the AK112-containing regimen was as long as 19.3 months. At the 2024 ESMO conference, a study on the safety and efficacy of AK112 combined with paclitaxel or albumin-bound paclitaxel as first-line treatment for advanced TNBC was reported. The study results showed that the overall ORR was 78.8%, the 6-month PFS rate was 73.3%, and the mPFS and OS have not yet been reached. These results suggest that AK112 may also have great application potential in TNBC patients with brain metastasis. In addition, sacituzumab govitecan is a novel ADC targeting TROP2. Based on the results of the large-scale phase III ASCENT study, it has been approved for the treatment of second-line and later-line metastatic TNBC. Through subgroup analysis of brain metastasis patients in the ASCENT study, we found that the PFS of brain metastasis patients in the SG group was significantly better than that of the control chemotherapy group (2.8 months vs. 1.6 months), indicating that ADCs targeting the TROP2 also have good efficacy in TNBC brain metastasis. Therefore, a prospective, single-arm, phase II clinical study of AK112 combined with TROP2 ADC in the treatment of triple-negative breast cancer brain metastasis is planned, aiming to explore the efficacy and safety of AK112 combined with TROP2 ADC in the treatment of TNBC brain metastasis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 70 years, with no gender restrictions;
2. ECOG performance score of 0 to 2;
3. Expected survival ≥ 3 months;
4. Patients with unresectable locally advanced, recurrent or metastatic triple-negative breast cancer who have failed treatment with taxane drugs are included.
5. Ten tissue pathology slides of the primary lesion and/or metastatic lesion (preferably metastatic lesion) can be obtained before the start of treatment for exploratory analysis of molecular indicators related to therapeutic efficacy.
6. Patients must have brain metastases confirmed by MRI, with at least one brain metastasis lesion that previously has not received radiotherapy and has a longest diameter of ≥ 1.0 cm; for brain metastasis lesions that have received local treatment, progression must be confirmed by imaging examination;
7. Cohort A: Patients with brain metastases who have not received central nervous system radiotherapy before. Patients with new brain lesions after craniotomy are allowed to be included, provided that they have not received radiotherapy after surgery and at least 2 weeks have passed since the surgery;
8. Cohort B: Patients with lesion progression or new lesions after whole brain radiotherapy (WBRT) or stereotactic radiotherapy (SRT). If a patient has multiple central nervous system lesions and only one or a few of them have received SRT treatment, and there are untreated lesions, such patients are still eligible for inclusion in this study;
9. The use of mannitol or hormones for treatment is allowed before enrollment, but the hormone treatment dose should be stable for at least one week without the need for an increase;
10. All patients enrolled are required to have adequate hematologic, hepatic, and renal function;
11. Be able to understand the study procedures and sign informed consent.

Exclusion Criteria:

1. Patients with soft meningeal metastases confirmed by MRI or lumbar puncture;
2. Presence of third-space effusion that cannot be controlled by drainage or other methods (such as large amounts of pleural effusion and ascites);
3. Received whole brain radiotherapy, chemotherapy, or surgery within 2 weeks before the treatment with the investigational drug, or received targeted therapy or endocrine therapy within 1 week before the treatment;
4. Previously used monoclonal or bispecific antibodies containing anti-VEGF-A and anti-PD-1/PD-L1/CTLA-4; previously used TROP2 ADC drugs.
5. Participated in other drug clinical trials within 2 weeks before enrollment;
6. Simultaneously receiving any anti-tumor treatment for other tumors;
7. Had other malignant tumors within the past 5 years, excluding cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinoma of the skin, differentiated thyroid cancer, etc. that have been cured;
8. Patients with severe heart diseases, including: (1) Congestive heart failure (NYHA class > 2); (2) History of unstable angina pectoris; (3) Myocardial infarction within the past 48 weeks; (4) Clinically significant arrhythmias (excluding atrial fibrillation and paroxysmal supraventricular tachycardia); (5) Any other heart diseases deemed by the investigator as unsuitable for participation in this trial;
9. Known hypersensitivity to the components of the investigational drug;
10. Uncontrolled serious infection.

10. History of immunodeficiency, including HIV positive, active hepatitis C virus infection or other acquired or congenital immunodeficiency diseases, or history of organ transplantation; patients with positive hepatitis B surface antigen (HBsAg) and HBV DNA > 2000 IU/ml or > 104 copies/ml should receive antiviral treatment according to local treatment guidelines and be willing to receive antiviral treatment throughout the study period; 11. Use of live attenuated vaccines within 28 days before randomization, or expected to use such vaccines during the study period (patients are not allowed to receive live attenuated influenza vaccine within 4 weeks before randomization, during treatment, and within 5 months after the last dose of SHR-1316/placebo); 12. Active, known or suspected autoimmune diseases, including but not limited to myasthenia gravis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, etc. Type 1 diabetes (controlled by insulin), hypothyroidism due to autoimmune thyroiditis that only requires hormone replacement therapy, or conditions that are not expected to recur without external stimulation are allowed. Patients with eczema, psoriasis, chronic simple lichen or only with skin manifestations of vitiligo (excluding psoriatic arthritis) can be enrolled if the rash covers less than 10% of the body surface area, the disease is well controlled at baseline and only requires low-potency topical steroids, and there has been no acute exacerbation of the underlying disease in the past 12 months (no need for psoralen plus ultraviolet radiation [PUVA], methotrexate, retinoids, biologics, oral calcineurin inhibitors, high-potency or oral steroids); 13. History of definite neurological or mental disorders, including epilepsy or dementia; 14. Pregnant or lactating women, women of childbearing age with positive baseline pregnancy test, or women who are unwilling to take effective contraceptive measures throughout the study period; 15. According to the investigator's judgment, patients with severe concomitant diseases that may endanger their safety or affect their completion of the study (including but not limited to uncontrolled severe hypertension, severe diabetes, active infection, thyroid disease, etc.); 16. Any other conditions deemed by the investigator as unsuitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Intracranial objective response rate (CNS ORR) | Up to approximately 12 weeks
  CNS ORR is the percentage of participants with the best objective response of complete response (CR) or partial response (PR) of Intracranial metastatic lesions according to RANO-BM criteria. CR = Disappearance of all non-nodal target lesions. PR = At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.

SECONDARY OUTCOMES:
Intracranial clinical benefit rate (CNS CBR) | Up to approximately 12 weeks
  Percentage of participants with complete response (CR) or partial response (PR) or stable disease (SD) lasting 4 weeks or longer of intracranial metastatic lesions as defined in RANO-BM criteria.
Progression-Free Survival (PFS) | Up to approximately 30 months
  PFS defined as the time from the date of randomization to the first evidence of disease progression as defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant does not have a complete baseline disease assessment, then the PFS time was censored at the date of randomization, regardless of whether or not objectively determined disease progression or death has been observed for the participant. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date.
Overall Survival (OS) | Up to approximately 30 months
  Time from date of randomization to the date of death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bardia A, Rugo HS, Tolaney SM, Loirat D, Punie K, Oliveira M, Brufsky A, Kalinsky K, Cortes J, Shaughnessy JO, Dieras V, Carey LA, Gianni L, Piccart-Gebhart M, Loibl S, Yoon OK, Pan Y, Hofsess S, Phan SC, Hurvitz SA. Final Results From the Randomized Phase III ASCENT Clinical Trial in Metastatic Triple-Negative Breast Cancer and Association of Outcomes by Human Epidermal Growth Factor Receptor 2 and Trophoblast Cell Surface Antigen 2 Expression. J Clin Oncol. 2024 May 20;42(15):1738-1744. doi: 10.1200/JCO.23.01409. Epub 2024 Feb 29. PMID 38422473
- [Background] Naito Y, Nakamura S, Kawaguchi-Sakita N, Ishida T, Nakayama T, Yamamoto Y, Masuda N, Matsumoto K, Kogawa T, Sudo K, Shimomura A, Lai C, Zhang D, Iwahori Y, Gary D, Huynh D, Iwata H. Preliminary results from ASCENT-J02: a phase 1/2 study of sacituzumab govitecan in Japanese patients with advanced solid tumors. Int J Clin Oncol. 2024 Nov;29(11):1684-1695. doi: 10.1007/s10147-024-02589-x. Epub 2024 Sep 20. PMID 39302614
- [Background] Frentzas S, Austria Mislang AR, Lemech C, Nagrial A, Underhill C, Wang W, Wang ZM, Li B, Xia Y, Coward JIG. Phase 1a dose escalation study of ivonescimab (AK112/SMT112), an anti-PD-1/VEGF-A bispecific antibody, in patients with advanced solid tumors. J Immunother Cancer. 2024 Apr 19;12(4):e008037. doi: 10.1136/jitc-2023-008037. PMID 38642937
- [Background] Zhao Y, Chen G, Chen J, Zhuang L, Du Y, Yu Q, Zhuang W, Zhao Y, Zhou M, Zhang W, Zhang Y, Wan Y, Li W, Song W, Wang ZM, Li B, Xia M, Yang Y, Fang W, Huang Y, Zhang L. AK112, a novel PD-1/VEGF bispecific antibody, in combination with chemotherapy in patients with advanced non-small cell lung cancer (NSCLC): an open-label, multicenter, phase II trial. EClinicalMedicine. 2023 Aug 3;62:102106. doi: 10.1016/j.eclinm.2023.102106. eCollection 2023 Aug. PMID 37593227